CLINICAL TRIAL: NCT06946992
Title: The Effect of Video Supported Cooperative Learning on Nursing Students' OSCE Achievement and Self-Efficacy Perceptions: A Randomized Controlled Study
Brief Title: The Effect of Video Supported Cooperative Learning
Acronym: OSCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Evrim Eyikara, Assistant professor, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: GaziU-HF-ES-03
Record Dates: First submitted 2025-04-12; First posted 2025-04-27 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-04

CONDITIONS: OSCE (Objective Structured Clinical Examination); Video-Assisted; Nursing Education
Keywords: cooperative learning; nursing education; nursing students; OSCE; video assisted

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- video supported cooperative learning (Experimental): Video supported cooperative learning will be used in the experimental group. The process will be student-centered. Students will be divided into groups of 8-10 students. Students will work on the psychomotor skills they are responsible for in the OSCE exam with cooperative learning method and in small groups on models. In this process, students will support each other's learning. They will reinforce their practices by watching the videos prepared for each psychomotor skill learning while practicing on the models in the form of cooperative learning.
  Interventions: Other: video supported cooperative learning
- traditional education (control group) (No Intervention): In the control group, educator-centered traditional laboratory practice will be carried out. Students will be divided into groups of 8-10 students. They will practice the psychomotor skills they are responsible for in the OSCE exam on the models with the help of the educator. In this process, an educator will be present next to each small group and will act as a guide.

INTERVENTIONS:
Other: video supported cooperative learning — Video supported cooperative learning will be used in the experimental group. The process will be student-centered. Students will support each other's learning. While practicing on the models in the form of cooperative learning, they will reinforce their practices by watching videos prepared for each psychomotor skill learning.
  Arms: video supported cooperative learning

SUMMARY:
This study will be conducted in a randomized controlled design to determine the effect of video-supported collaborative learning on nursing students' OSCE achievement and self-efficacy perceptions. The research population will consist of first-year nursing students enrolled in the Nursing principles course (n = 24). A research group consisting of 100 participants is planned. Considering the inclusion criteria, students who volunteered to participate in the study will be identified. "Descriptive characteristics form" and 'Brief and Universal Self-Efficacy Scale for Clinical Skills' (pre-test) will be administered to the students. Students will be randomized according to their mean scores on the scale and experimental and control groups will be formed. . Students will take the OSCE exam at the end of the spring semester. For the preparation of OSCE, free laboratory studies are organized beforehand. Video supported cooperative learning will be used in the experimental group. The process will be student-centered. In the control group, educator-centered traditional laboratory practice will be used. After 16 hours of free laboratory work, the "Brief and Universal Self-Efficacy Scale for Clinical Skills" (post-test) will be administered to all students in the sample group. One week after the free laboratory work, OSCE exam will be conducted. While the students perform the skill steps, the trainers will mark one of the options 'correct', 'incorrect or incomplete', 'not observed' for each step on the OSCE checklist.

DETAILED DESCRIPTION:
Teaching methods used in nursing education have changed differently from past to present. Today, technology-supported teaching methods have become widespread. Today's students are self-learners who use technology well, like to learn with technological tools and equipment. These students prefer to learn by taking advantage of the conveniences provided by technology.

One of the approaches used in psychomotor skill assessment is the Objective Structured Clinical Examination (OSCE). In OSCE, which enables direct assessment of various clinical skills, a "station" is prepared for each skill to be assessed. The skill performances and competencies of the students at each station are evaluated by the educators. The use of structured checklists in skill assessment ensures that each student is evaluated objectively.

One of the most frequently preferred technologies in the literature recently to improve nursing students' OSCE achievement and self-efficacy perceptions is skill videos and collaborative learning.

In this context, this study will be conducted in a randomized controlled design to determine the effect of video-supported collaborative learning on nursing students' OSCE achievement and self-efficacy perceptions.

The population of the study will consist of first-year nursing students (n=243) enrolled in the Nursing Principles course at Gazi University Faculty of Nursing in the spring semester of the 2024-2025 academic year. Students who volunteered to participate in the study and met the inclusion criteria will constitute the sample group. Power analysis was performed in GPower 3.1.9.7 program to determine the sample size. In order to determine the difference between the groups in terms of measurements, 45 people in the groups were determined as 90 people in total according to type 1 error: 0.05 type 2 error: 0.20 and effect size= 0.60. Considering the calculated situation due to possible losses in the study, the sample size was increased by 10% and it was planned to take 100 people, 50 in groups.

"Descriptive characteristics form" and 'Brief and Universal Self-Efficacy Scale for Clinical Skills' (pre-test) will be administered to all students. Then, students who volunteered to participate in the study will be determined by considering the inclusion criteria. Students will be randomized according to their mean scores on the scale and experimental and control groups will be formed.

Students will take the OSCE exam at the end of the spring semester of the 2024-2025 academic year. For the preparation of OSCE, free laboratory studies are organized beforehand. Students in the experimental and control groups will perform psychomotor skill practices before OSCE using a different teaching method. However, the training of the groups will be carried out in different laboratories and simultaneously:

Video supported cooperative learning will be used in the experimental group. The process will be student-centered. Students will be divided into groups of 8-10 students. Students will work on the psychomotor skills they are responsible for in the OSCE exam with cooperative learning method and in small groups on models. In this process, students will support each other's learning. While practicing on the models in the form of cooperative learning, they will reinforce their practices by watching videos prepared for each psychomotor skill learning. In this process, an educator will be present with each small group and will assume a facilitating role. He/she will correct students if they are wrong/deficient and support learning.

In the control group, educator-centered traditional laboratory practice will be carried out. Students will be divided into groups of 8-10 students. They will practice the psychomotor skills they are responsible for in the OSCE exam on the models with the help of the educator. In this process, an educator will be present with each small group and will act as a guide. He/she will correct students' mistakes and support learning. Videos prepared for each psychomotor skill learning will be given to the students in advance and they will be asked to watch them.

After 16 hours of free laboratory work, the "Brief and Universal Self-Efficacy Scale for Clinical Skills" (post-test) will be administered to all students in the sample group. One week after the free laboratory work, the OSCE exam will be conducted. Each student will be given approximately 7-8 minutes at each station to complete the skill steps. Experimental and control group students will take the OSCE on the same day on the same basic nursing skills. While the students are performing the skill steps, the trainers will mark one of the options 'correct', 'incorrect or incomplete', 'not observed' for each step on the OSCE checklist. The week after the OSCE, the control group and the students who were not included in the study will be given the opportunity for free laboratory work accompanied by a video so that everyone can benefit equally. These procedures will end in the spring semester of the academic year.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in the Nursing Principles course for the first time,
* participation in the laboratory practices of the Nursing Principles course
* volunteering to participate in the study.

Exclusion Criteria:

* High school, associate degree or bachelor's degree in a health-related field,
* Difficulty speaking and understanding Turkish.
* Removal criteria from the study (If the student wants to leave the study at any stage and does not fill in the data collection forms)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2025-04-30 (Actual); Primary Completion 2025-05-23 (Actual); Study Completion 2025-05-23 (Actual)

PRIMARY OUTCOMES:
Brief and Universal Self-Efficacy Scale for Clinical Skills | an average of four weeks from baseline to study completion
  The scale was developed by Kang et al. in 2019 to measure students' self-efficacy perception towards tasks requiring skills (professional skills for practice) and Turkish validity and reliability study was conducted by Bayazıt et al. (2022). As a result of Turkish validity and reliability, Cronbach Alpha internal consistency coefficient was found to be 0.91. The scale is a Likert-type scale consisting of 15 items and 3 sub-dimensions scored between 1-5. The lowest score is 18 and the highest score is 90. The high score obtained from each sub-dimension of the scale indicates that the individual has the characteristic evaluated by the relevant sub-dimension.
OSCE checklists | once the study is completed, at the end of 4 weeks
  The checklist was prepared by the researchers and in line with the literature. The first checklist includes "drug administration and fluid requirement", the second checklist includes "nasopharyngeal/tracheal aspiration" and the third checklist includes "enema administration and intermittent feeding with nasogastric catheter". It consists of practice steps that question psychomotor skill steps in detail. It was created in the form of a rubric for objective observation of the students. Expert opinions will be taken and the content validity index will be calculated. The total score to be obtained from the entire checklist is 150.

CONTACTS AND LOCATIONS:
Overall Officials: Evrim EYİKARA SARITAŞ, Principal Investigator — Gazi University
Locations (1):
- Gazi University Faculty of Nursing, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No